CLINICAL TRIAL: NCT02788812
Title: The Comparison of the Quality of Life and Outcomes in Patient's With Incarcerated Inguinal Hernias: Laparoscopic Transabdominal Pre-peritoneal (TAPP) Versus Modified Lichtenstein Hernioplasty
Brief Title: QOL in Incarcerated Inguinal Hernias: TAPP Vs Open Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarawak General Hospital (Other)
Responsible Party: Principal Investigator, Siow Sze Li, Dr, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-16-453-29942
Record Dates: First submitted 2016-05-21; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open modified Lichtenstein repair (Active Comparator)
  Interventions: Procedure: Open modified Lichtenstein repair
- Laparoscopic TAPP inguinal hernia repair (Active Comparator)
  Interventions: Procedure: Laparoscopic TAPP inguinal hernia repair

INTERVENTIONS:
Procedure: Open modified Lichtenstein repair — Open Lichtenstein Hernioplasty
  Arms: Open modified Lichtenstein repair
Procedure: Laparoscopic TAPP inguinal hernia repair — Laparoscopic TAPP Hernioplasty
  Arms: Laparoscopic TAPP inguinal hernia repair

SUMMARY:
To determine if there is a difference in the quality of life in between patients who undergoes laparoscopic transabdominal pre-peritoneal (TAPP) or modified Lichtenstein hernioplasty

DETAILED DESCRIPTION:
Patients presenting with incarcerated inguinal hernias will be randomized between open or laparoscopic repair groups. The primary outcome will be the quality of life scores. Patients will be followed-up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Both genders
* Unilateral inguinal hernias
* Incarcerated inguinal hernias
* Elective setting

Exclusion Criteria:

* Anaesthesiologists) Grade > 2
* Recurrence
* Inguinal-scrotal hernias
* Prostatectomy, Pfannenstiel incision, previous pre-peritoneal surgery
* Pregnancy
* Refusal for general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores as measured by Carolinas Comfort Scale | 12 months
  Carolina Comfort Scale during the duration of follow-up

SECONDARY OUTCOMES:
Operating Time in Minutes | 12 months
  Comparing the duration of operation between open and laparoscopic surgeries.
Duration of Hospitalization in Days | 12 months
  Comparing the duration of post operative stay between open and laparoscopic surgeries.
Recurrence of Hernia after Operation | 12 monthts
  Comparing the recurrences between open and laparoscopic surgeries.

IPD SHARING:
Plan to Share IPD: No